CLINICAL TRIAL: NCT00777322
Title: Pilot Study of Excimer Laser Topography-Computer Assisted Treatment (T-Cat) Combined With Corneal Collagen Cross-linking With Riboflavin and UV Light
Brief Title: T-Cat Laser & Cross-linking for Keratoconus
Acronym: T-Cat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Accuvision Laser Eye Clinics (Other); Carleton Optical Equipment Ltd. (Industry); Bon Optics (Other); Sooft Italia (Industry)
Responsible Party: Mr Chad K Rostron, Moorfields Eye Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC Ref: 07/H0721/94
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2009-04

CONDITIONS: Keratoconus; Pellucid Marginal Degeneration
Keywords: keratoconus; pellucid marginal degeneration; corneal ectasia; collagen cross-linking; riboflavin; UV light; excimer laser; Topography-Computer Assisted Treatment (T-Cat); Wavelight Allegretto laser
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin; Dextrans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional study (Experimental): Patients with known keratoconus or pellucid marginal degeneration will be invited to join the study. The study is partly a continuation in the management of patients who have had previous keratophakia, who will have near-normal or supra-physiological levels of corneal thickness. It is also intended for patients with relatively mild keratoconus who have sufficient corneal thickness to allow a limited laser ablation whilst still leaving a residual stromal bed of at least 350μ.
  Interventions: Procedure: Excimer laser ablation, and collagen cross-linking

INTERVENTIONS:
Procedure: Excimer laser ablation, and collagen cross-linking — Surgery is performed with topical anaesthesia. The central corneal epithelium is removed. Excimer laser ablation is applied (typically 15-30 seconds). Residual bed thickness is checked with an ultrasonic pachymeter. Topical application of riboflavin 0.1% in dextran is commenced at 5 minute intervals. When an adequate saturation of the anterior chamber with riboflavin has been achieved, cross-linking treatment will proceed. Output from the UV light generating equipment is measured with a UV light meter and set at 3mW/cm². Thirty minutes of treatment is given, interrupted at five minute intervals by the application of more topical riboflavin drops. Finally the eye has a bandage soft contact lens placed, with preservative free topical antibiotic, steroid, and cycloplegic drop application.
  Other Names: Ricrolin (riboflavin 0.1% in dextran); Pecshke UV-X illumination system

SUMMARY:
The purpose of this study is to determine whether excimer laser corneal surface ablation (T-Cat) can be safely combined with simultaneous corneal collagen cross-linking treatment to produce an improved and stable corneal profile in the treatment of keratoconus.

DETAILED DESCRIPTION:
Theoretical framework:

Corneal ectasia is a relative weakness in the structure of the cornea, which produces a progressive change in its shape with resultant visual distortion.

Excimer laser surface ablation can be used to re-shape the corneal profile. When the corneal shape is very irregular, corneal topography data gives the best information as to how to re-shape the cornea into a normal profile, and this Topography-Computer Assisted Treatment (T-Cat) will be used to modulate the surface corneal shape.

It is known that collagen cross-linking in the cornea occurs naturally with age, and in diabetes, both of which seem to prevent progressive ectasia. Corneal collagen cross-linking with riboflavin has been shown to stabilize the cornea in keratoconus, and prevents progression of the disease. If cross-linking is performed at that moment that the cornea has been re-shaped by T-Cat treatment, it should help prevent the corneal thinning resultant from the laser treatment from destabilising the cornea and causing progressive ectasia.

Purpose:

To determine whether excimer laser corneal surface ablation (T-Cat) can be safely combined with simultaneous corneal collagen cross-linking treatment to produce an improved and stable corneal profile.

Design:

Prospective, interventional trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known keratoconus or pellucid marginal degeneration.

Exclusion Criteria:

* Age < 18 years > 50 years.
* Minimal corneal pachymetry in eye to be treated of < 400μ.
* Evidence of other corneal disease in the eye to be treated (e.g. Herpes simplex keratitis).
* Women who are pregnant or nursing at the time of the initial treatment.
* Presence of significant central corneal opacity.
* Patients unwilling to not wear rigid contact lenses in the eye to be operated on for at least one month before baseline examination, and for the first six months post-operatively.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The difference in the pre- and post-operative unaided visual acuity, best corrected visual acuity, and refraction. | At six months

SECONDARY OUTCOMES:
Corneal topographic profile. | At six months

CONTACTS AND LOCATIONS:
Overall Officials: Chad K Rostron, MB BS, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Department at St George's Hospital, London, London, United Kingdom